CLINICAL TRIAL: NCT03071380
Title: Comparative Randomized, Single Dose, Two-way Crossover Open-label Study to Determine the Bioequivalence of Rivaroxaban From Repatoxaban 10 mg Tablets (Horus for Pharmaceutical Industries, Egypt) and Xarelto® 10 mg Tablets (Janssen Pharm., Licensed From: Bayer Healthcare, Germany)
Brief Title: Bioequivalence Study of Rivaroxaban From Repatoxaban 10 mg Tablets (Horus for Pharmaceutical Industries, Egypt) and Xarelto® 10 mg Tablets (Janssen Pharm., Licensed From: Bayer Healthcare, Germany)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genuine Research Center, Egypt (Industry)
Collaborators: Horus for Pharmaceutical Industries, Egypt (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GRC/1/14/548
Record Dates: First submitted 2017-03-01; First posted 2017-03-06 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Healthy
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- T test (Experimental): Test drug (Repatoxaban) 1 tablet contains 10 mg rivaroxaban
  Interventions: Drug: Repatoxaban
- B reference (Active Comparator): Reference drug (Xarelto) 1 tablet contains 0 mg rivaroxaban
  Interventions: Drug: Xarelto

INTERVENTIONS:
Drug: Repatoxaban — 1 tablet contains 10 mg rivaroxaban
  Other Names: Xarelto
  Arms: T test
Drug: Xarelto — 1 tablet contains 10 mg rivaroxaban
  Arms: B reference

SUMMARY:
An open label randomized, single dose, two-way crossover bioequivalence study to determine the bioequivalence of Rivaroxaban from Repatoxaban 10 mg Tablets (Horus for Pharmaceutical Industries, Egypt) and Xarelto® 10 mg Tablets (Janssen Pharm., Licensed from: Bayer Healthcare, Germany)

DETAILED DESCRIPTION:
Primary Pharmacokinetic Parameters: Cmax, AUC0→t and AUC0→∞ Secondary Pharmacokinetic Parameters: Ke, tmax and t1/2e. ANOVA using 5% significance level for transformed (with the 90% confidence intervals) and untransformed data of Cmax, AUC0→t and AUC0→∞ and for untransformed data of Ke, tmax and t1/2e.

The confidence intervals of logarithmically transformed Test/Reference ratios for Cmax, AUC0→t and AUC0→∞ to be within 80.00-125.00%.

A comprehensive final report will be issued upon the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, age 18 to 55 years, inclusive.
2. Body weight within 15% of normal range according to the accepted normal values for body mass index (BMI).
3. Medical demographics without evidence of clinically significant deviation from normal medical condition.
4. Results of clinical laboratory test are within the normal range or with a deviation that is not considered clinically significant by principal investigator.
5. Subject does not have allergy to the drugs under investigation.

Exclusion Criteria:

1. Subjects with known allergy to the products tested.
2. Subjects whose values of BMI were outside the accepted normal ranges.
3. Female subjects who were pregnant, nursing or taking birth control pills.
4. Medical demographics with evidence of clinically significant deviation from normal medical condition.
5. Results of laboratory tests which are clinically significant.
6. Acute infection within one week preceding first study drug administration.
7. History of drug or alcohol abuse.
8. Subject does not agree not to take any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.
9. Subject is on a special diet (for example subject is vegetarian).
10. Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.
11. Subject does not agree not to consume any beverages or foods containing grapefruit 7 days prior to first study drug administration until the end of the study.
12. Subject has a history of severe diseases which have direct impact on the study.
13. Participation in a bioequivalence study or in a clinical study within the last 6 weeks before first study drug administration.
14. Subject intends to be hospitalized within 3 months after first study drug administration.
15. Subjects who, through completion of this study, would have donated more than 500 ml of blood in 7 days, or 750 ml of blood in 30 days, 1000 ml in 90 days, 1250 ml in 120 days, 1500 ml in 180 days, 2000 ml in 270 days, 2500 ml of blood in 1 year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Maximal measured plasma concentration (Cmax) | Up to 48 hours post dose in each treatment period
  Serial blood samples for determination of study drug will be collected at 0.00, 0.33, 0.66, 1.00, 1.50, 2.00, 2.50, 3.00, 3.5, 4.00, 6.00, 8.00, 12.00, 24.00 and 48.00 hours

SECONDARY OUTCOMES:
Time of the maximum plasma concentration (Tmax) | Up to 48 hours post dose in each treatment period
  The amount of time that a drug is present at the maximum concentration in serum

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshafeey, Ph.D. Pharma, Study Director — Genuine Research Center
Locations (1):
- Genuine Research Center GRC, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chow SC, Wang H. On sample size calculation in bioequivalence trials. J Pharmacokinet Pharmacodyn. 2001 Apr;28(2):155-69. doi: 10.1023/a:1011503032353. PMID 11381568
- [Background] Diletti E, Hauschke D, Steinijans VW. Sample size determination for bioequivalence assessment by means of confidence intervals. Int J Clin Pharmacol Ther Toxicol. 1991 Jan;29(1):1-8. PMID 2004861
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848